CLINICAL TRIAL: NCT04743947
Title: Observational Study on the Effects of SARS-CoV-2 Vaccination in Dialysis and Kidney Transplant Patients
Brief Title: Vaccination Against COVID-19 in Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, PD Dr. med. Johannes Stegbauer, Assistant Professor, Heinrich-Heine University, Duesseldorf
Other Study IDs: 2020-1237
Record Dates: First submitted 2021-02-04; First posted 2021-02-08 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Chronic Kidney Disease Stage 5 on Dialysis; Chronic Kidney Disease Stage 5 With Transplant; Vaccine Response Impaired
Keywords: SARS-CoV-2; vaccination; dialysis; kidney transplantation
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with kidney failure receiving dialysis: Analysis of data received from clinical practice about the SARS-CoV-2 vaccination response in dialysis patients (hemodialysis or peritoneal dialysis).
  Interventions: Other: No intervention; observational study
- Kidney transplant patients: Analysis of data received from clinical practice about the SARS-CoV-2 vaccination response in kidney transplant patients.
  Interventions: Other: No intervention; observational study
- age-matched controls in non-dialysis, non-kidney transplant patients: Historical cohort of aged matched non-dialysis and non-kidney transplanted patients who received a SARS-CoV-2 vaccination.
  Interventions: Other: No intervention; observational study

INTERVENTIONS:
Other: No intervention; observational study — no intervention

SUMMARY:
This is a prospective, multi-center, observational study that will enroll patients receiving dialysis (hemodialysis or peritoneal dialysis) or patients with kidney transplantation who will be vaccinated against COVID-19.

DETAILED DESCRIPTION:
Patients on dialysis and kidney transplant patients infected with SARS-CoV-2 (severe acute respiratory syndrome coronavirus type 2) have an increased risk to develop a more severe course of disease or die from COVID-19 (coronavirus disease 2019). SARS-CoV-2 vaccination can increase protection against COVID-19. Kidney transplant patients and patients requiring dialysis suffer from an acquired immune deficiency. Due to the dysfunctional immune response, the general vaccine response in dialysis patients and kidney transplant patients is in many cases insufficient.

Until now, the vaccination response in dialysis patients and kidney-transplanted patients is unpredictable. Verification of vaccine response can provide important information on how to treat and protect these patients from a COVID-19. Therefore, there is a medical need to monitor vaccine protection after SARS-CoV-2 vaccination in clinical practice. In this observational study, data of the SARS-CoV-2 vaccination response collected in clinical routine will be analyzed from these patients. Based on this observational study, the investigators aim to get first evidence whether and to what extent vaccination against COVID-19 causes a vaccine response in immunocompromised patients with kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* receiving dialysis (hemodialysis or peritoneal dialysis)
* capable of giving consent
* age 18 or older

Exclusion Criteria:

- non-capable of giving consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated in a nephrology in- or out-patient clinic and how are willing to get a SARS-CoV-2 vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2- antibody- titer | 2 years
  SARS-CoV-2- antibody- titer after vaccine

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - MVZ DaVita Rhein-Ruhr, Düsseldorf
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Düsseldorf
  - University Hospital Düsseldorf, Heinrich Heine University, Düsseldorf
  - Nephrocare Mettmann, Mettmann
  - Hospital Solingen, Solingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kolb T, Fischer S, Muller L, Lubke N, Hillebrandt J, Andree M, Schmitz M, Schmidt C, Kucukkoylu S, Koster L, Kittel M, Weiland L, Dreyling KW, Hetzel G, Adams O, Schaal H, Ivens K, Rump LC, Timm J, Stegbauer J. Impaired Immune Response to SARS-CoV-2 Vaccination in Dialysis Patients and in Kidney Transplant Recipients. Kidney360. 2021 Jul 13;2(9):1491-1498. doi: 10.34067/KID.0003512021. eCollection 2021 Sep 30. PMID 35373105